CLINICAL TRIAL: NCT07338552
Title: A Virtual Community-Based Digital Intervention for Prediabetes Management in China
Brief Title: Effectiveness of a Virtual Health Management Community (VHMC) for Pre-diabetes in China
Acronym: VHMC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiling Hu, Chief Nurse, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RG2023-262-02; 72204277 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-12-19; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Prediabetes
Keywords: Prediabetes; Health management
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Other: Usual Care
- Intervention Group (Experimental)
  Interventions: Behavioral: VHMC-based Group Interaction Management

INTERVENTIONS:
Other: Usual Care — The control group participants will receive conventional health education including disease-related knowledge, diet skills, exercise skills, comprehensive management goals (for blood glucose, weight, blood pressure, and blood lipids), and general education regarding lifestyle modification, delivered verbally or in the form of pamphlets.
  Arms: Control group
Behavioral: VHMC-based Group Interaction Management — The intervention group will receive group interaction management based on the Virtual Health Management Community (VHMC) plan. After enrollment, health managers and patients will participate in face-to-face group consultations to clarify roles and responsibilities in self-management and group management, elicit patients' self-motivation statements, and jointly develop meaningful individual- and group-level goals. Health managers will then assist patients in downloading the VHMC platform application and guide them through its modules. After the face-to-face consultations, patients will log into the platform at home to access health information, record diabetes-related daily experiences, participate in community interactions, and implement lifestyle interventions. Health managers will continuously assess participants' progress in knowledge acquisition and lifestyle implementation and provide feedback and guidance throughout the intervention period.
  Arms: Intervention Group

SUMMARY:
Individuals with prediabetes are at high risk for developing type 2 diabetes mellitus (T2DM) and are therefore prone to serious complications such as stroke, kidney failure, blindness, and lower-limb amputation. Prediabetes can be reversed, and lifestyle modification is considered the most effective intervention for diabetes prevention. However, it is difficult for individuals with prediabetes to maintain long-term healthy lifestyle changes owing to psychological burnout and poor adherence during daily self-management. We developed a novel virtual health management community (VHMC) model based on group interaction management. The purpose of this study is to evaluate whether a virtual health management community-based intervention can improve glycemic control and related health outcomes in adults with prediabetes.

Participants in the intervention group will receive lifestyle management support through a virtual health management community, including health education, lifestyle guidance, and group-based interaction delivered via a digital platform.

Participants will be randomly assigned to either the virtual health management community intervention group or a usual care control group.

The study will follow participants for approximately 6 months.

Participants in the intervention group will receive lifestyle management support through a virtual health management community, including health education, lifestyle guidance, and group-based interaction delivered via a digital platform.

Participants will be randomly assigned to either the virtual health management community intervention group or a usual care control group.

The study will follow participants for approximately 6 months.

DETAILED DESCRIPTION:
Prediabetes, including impaired fasting glucose (IFG) and impaired glucose tolerance (IGT), is a metabolic state characterized by elevated blood glucose levels that do not yet meet the diagnostic criteria for diabetes. China has the highest prevalence of prediabetes among adults, estimated at 35.2%. Individuals with prediabetes are at high risk of progressing to type 2 diabetes mellitus (T2DM), which is associated with severe complications such as cardiovascular disease, kidney failure, blindness, and substantial economic burden. Therefore, preventing the progression from prediabetes to diabetes is an urgent public health priority.

Lifestyle modification is recognized as the most effective strategy for diabetes prevention; however, long-term adherence remains challenging. Traditional self-management interventions predominantly focus on individual-level behavior change, often overlooking the role of social support and community engagement. Group-based health management has the potential to provide social, practical, and emotional support, thereby enhancing self-efficacy, but existing models are frequently passive, fragmented, and difficult to sustain over time.

Virtual health communities (VHCs) provide online platforms that facilitate social interaction and self-management, overcoming geographical and time constraints while promoting active engagement. Although VHC-based group management approaches have been applied in various chronic diseases, their application in individuals with prediabetes remains limited. Moreover, many existing models lack sufficient group interaction and emotional engagement to support sustained behavior change.

To address these gaps, we developed a novel Virtual Health Management Community (VHMC) model that integrates structured group interaction management with digital health support, including dedicated patient and health manager modules. This study aims to apply the VHMC platform in individuals with prediabetes and to evaluate the effectiveness of this group interaction-based management model in improving glycemic control and related health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet the 1999 World Health Organization (WHO) diagnostic criteria and the 2010 American Diabetes Association (ADA) definition for prediabetes, including: impaired fasting glucose (IFG): fasting plasma glucose (FPG) 6.1-<7.0 mmol/L and 2-hour plasma glucose (2-hPG) <7.8 mmol/L during a 75-g oral glucose tolerance test (OGTT); or impaired glucose tolerance (IGT): FPG <7.0 mmol/L and 2-hPG 7.8-<11.1 mmol/L during a 75-g OGTT; or HbA1c 5.7%-6.4%;
* Age ≥18 years;
* Clear consciousness and adequate comprehension ability;
* Able to use a smartphone and have access to the Internet at home;
* Willing to participate in the study and provide written informed consent;
* Able to understand the purpose, procedure, and nature of the study.

Exclusion Criteria:

* Participants with significant cognitive impairment or mental disorders;
* Participants with severe malignant tumours;
* Participants with severe acute or chronic complications, such as blindness, heart failure, or end-stage renal disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Abnormal 2-hPG (OGTT; ≥11.1 mmol/L). | From enrollment to the end of intervention at 6 months

SECONDARY OUTCOMES:
HbA1c | From enrollment to the end of intervention at 6 months
Waist circumference | From enrollment to the end of intervention at 6 months
Hip circumferences | From enrollment to the end of intervention at 6 months
BMI | From enrollment to the end of intervention at 6 months
Dietary compliance assessed by the Food Frequency Questionnaire (FFQ) | From enrollment to the end of intervention at 6 months
Physical activity compliance assessed by the International Physical Activity Questionnaire (IPAQ) | From enrollment to the end of intervention at 6 months
Self-efficacy assessed by the General Self-Efficacy Scale (GSES) | From enrollment to the end of intervention at 6 months
Social support assessed by the Social Support Rating Scale (SSRS) | From enrollment to the end of intervention at 6 months
Illness perception assessed by the Brief Illness Perception Questionnaire (BIPQ) | From enrollment to the end of intervention at 6 months
Sense of coherence assessed by the 13-item Sense of Coherence scale (SOC-13) | From enrollment to the end of intervention at 6 months

IPD SHARING:
Plan to Share IPD: No
Due to participant privacy and confidentiality concerns, individual participant data will not be shared.